CLINICAL TRIAL: NCT04791787
Title: Effect of Ketogenic Diet on Glucose Metabolism and Energy Expenditure in Type 2 Diabetes CTMS 20-0042
Brief Title: Effect of Ketogenic Diet on Glucose Metabolism and Energy Expenditure in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20200230H
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Energy Supply; Deficiency; Type 2 Diabetes
Keywords: Ketogenic diet; Body fat; Insulin secretion
MeSH Terms: conditions — Glucose Metabolism Disorders; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into 3 groups. Each group will be assigned to one of 4 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Weight Maintenance (Active Comparator): Standard weight maintenance diet will be provided for 10 days for subjects who are not currently treated with a T2DM medication.
  Interventions: Other: Standard weight maintaining diet
- Isocaloric Diet (Active Comparator): Isocaloric diet will be provided for 10 days for subjects who are currently treated with a T2DM medication included in the inclusion criteria
  Interventions: Other: Weight maintaining isocaloric ketogenic diet
- Isocaloric Diet with Beta-hydroxy butyrate (Active Comparator): Isocaloric diet with Beta-hydroxy butyrate will be provided for 10 days for subjects who are not currently treated with a T2DM medication.
  Interventions: Other: Weight maintaining isocaloric ketogenic diet; Dietary Supplement: Beta-hydroxy butyrate

INTERVENTIONS:
Other: Standard weight maintaining diet — Diet containing diet approximately 25-35% protein, 45-55% carbohydrate, 20- 30% fat
  Arms: Standard Weight Maintenance
Other: Weight maintaining isocaloric ketogenic diet — Isocaloric ketogenic diet containing approximately 15-25% protein, 5-10% carbohydrate,70- 80% fat
  Arms: Isocaloric Diet; Isocaloric Diet with Beta-hydroxy butyrate
Dietary Supplement: Beta-hydroxy butyrate — A supplement of ketone ester of beta-hydroxy butyrate
  Other Names: BHOB
  Arms: Isocaloric Diet with Beta-hydroxy butyrate

SUMMARY:
The study team will examine the effect of a ketogenic diet alone and ketogenic diet supplemented with oral ketones on how the body of individuals with type 2 diabetes respond to insulin, regulates insulin secretion, food intake and energetic pathways and influences body fat distribution.

DETAILED DESCRIPTION:
Subjects will be randomized into three groups (1) standard, weight maintaining diet containing approximately 25-35% protein, 45-55% carbohydrate, 20-30% fat; (2) weight maintaining isocaloric ketogenic diet containing approximately 15-25% protein, 5-10% carbohydrate, 70-80% fat; (3) weight maintaining isocaloric diet containing approximately 15-25% protein, 5-10% carbohydrate, 70-80% fat supplemented with the ketone ester of beta-hydroxy butyrate, 8 grams every 8 hours to further increase the plasma ketone concentration by ~3 mM. Subjects will be further randomized on the basis of:

(i) HbA1c 7.0-8.5% and 8.5-10.5% to ensure similar baseline levels of glucose control and (ii) drug naïve versus drug-treated. At the time of screening, after a 10-12 hour overnight fast, indirect calorimetry will be performed with a ventilated hood system for 60 minutes to measure baseline energy expenditure. An initial weight maintenance energy requirement estimate as 1.5 times resting energy expenditure (obtained by indirect calorimetry) will be started. Diets will consist of a 10-day rotating menu using NutriAdmin for meal planning and Nutrition Maker for analysis of recipes Food will be prepared in the Cafeteria and or the Metabolic Kitchen at the Texas Diabetes Institute and certified by a dietician. Subjects will report to the diet kitchen at 8 AM on Monday through Saturday where they will eat their breakfast and pick up food for their lunch and dinner. On Saturday, participants also will be given food for their Sunday meals. Subjects will maintain a daily dietary log with all food consumed. On each visit subjects will be weighed; dietary log will be reviewed and the caloric content of the diet will be adjusted to maintain the body weight constant. Blood pressure will be measured in the reclining position x 2 separate days. Antidiabetic medications will not be changed during the study unless hypoglycemia (fasting plasma glucose <70 mg/dl or symptoms) occurs. The study duration will be 10 days which should be sufficient to observe the effect of hyperketonemia on glucose/lipid metabolism and energy expenditure. If participant cannot come on the last days of his/her diet treatment, than we will extend this period up to 13 days and participant will be given diet for additional days till completion of the study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-70 years
2. BMI = 27.5-42 kg.m2
3. HbA1c = 7.0-10.5
4. Weight stable (±4-5lb) in the preceding 3 months
5. Good general health

Exclusion Criteria:

1. Use of medications that affect glucose tolerance other than metformin/sulfonylurea/DPP4 Inhibitor
2. Major organ disease
3. Estimated Glomerular filtration rate (eGFR) <60 ml/min
4. Type 1 diabetes
5. Hematocrit < 34 (if HbA1c is in the 8.5 to 10% range)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) | Baseline to 10 days
  A change in FPG will be measured
Hepatic Glucose production (HGP) | Baseline to 10 days
  Change of hepatic glucose production will be measured using 3H-glucose infusion
Whole Body Fat Oxidation | Baseline to 10 days
  Change in whole body fat oxidation will be measured using indirect calorimetry
Total Body Fat | Baseline to 10 days
  Change in whole body fat
Hepatic Fat Content | Baseline to 10 days
  Change in hepatic fat content

SECONDARY OUTCOMES:
Plasma Insulin | Baseline to 10 days
  Change in plasma insulin will be measured
C-peptide | Baseline to 10 days
  Change in C-peptide will be measured
Free Fatty Acid (FFA) | Baseline to 10 days
  Change in FFA will be measured
Glycerol level | Baseline to 10 days
  Change in Glycerol level will be measured
Low density lipoproteins (LDL) | Baseline to 10 days
  Change in LDL
High density lipoproteins (HDL) | Baseline to 10 days
  Change in HDL
Triglycerides | Baseline to 10 days
  Change in triglyceride levels
Urine Microalbumin excretion | Baseline to 10 days
  Change in urine microalbumin excretion
Glycated hemoglobin test (HbA1c) | Baseline to 10 days
  Change in HbA1c
Fructosamine level | Baseline to 10 days
  Change in fructosamine

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (2):
- United States (2):
  - University Health Systems-Texas Diabetes Institute, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Information will be shared as summary results on ClinicalTrials.gov and in a peer-reviewed scientific journal publication
Supporting Information: Study Protocol, SAP
Time Frame: After study completion